CLINICAL TRIAL: NCT05700318
Title: A Pilot Study Assessing Preliminary Safety and Efficacy of The ShiraTronics Migraine Therapy System in Relieving, Interrupting, and Preventing Chronic Migraine
Brief Title: Study Using the ShiraTronics Migraine Therapy System
Acronym: RELIEV-CM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ShiraTronics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STCM01
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Chronic Migraine, Headache
MeSH Terms: conditions — Headache | interventions — Implantable Neurostimulators

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Neurostimulation (Experimental): Neurostimulation will be delivered to target nerves.
  Interventions: Device: neurostimulator

INTERVENTIONS:
Device: neurostimulator — The ShiraTronics Migraine Therapy System

SUMMARY:
The purpose of this pilot study is to assess the preliminary safety and efficacy of the ShiraTronics Migraine Therapy System in prophylactic treatment of patients with refractory chronic migraine.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who are 22 years of age or older.
2. History of migraine ≥ 12 months.
3. Participants experiencing between 15 to 26 headache days per month, with at least 8 headache days (per month) with migraine phenotype presentation.
4. Inadequate response to, unwilling, or contraindicated to Onabotulinumtoxin A and CGRP monoclonal antibodies therapy.
5. Stable use of migraine medication.

Exclusion Criteria:

1. Post-traumatic headache.
2. Medication overuse headache.
3. New daily persistent headache.
4. Report experiencing unremitting, continuous headaches with no relief.
5. Previously implanted neurostimulator to treat headache.
6. History of cervical radiofrequency ablation or had any other intervention/device for migraine.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Monthly Headache Days | 12-weeks
  Change in number of mean monthly headache days

SECONDARY OUTCOMES:
50% reduction in mean Headache days | 12-weeks
  Proportion of subjects with 50% reduction in mean monthly headache days
Monthly Migraine Days | 12-weeks
  Change in mean monthly migraine days
Migraine Disability Assessment Test | 12-weeks
  Change in disability score
Patient-identified Most Bothersome Symptom | 12-weeks
  Change in most bothersome symptom

CONTACTS AND LOCATIONS:
Overall Officials: Scientific Advisory Board, Study Director — ShiraTronics
Locations (4):
- Australia (4):
  - Genesis Research Services, Broadmeadow, New South Wales
  - Australian Medical Research, Hurstville, New South Wales
  - CerCare, Wayville, South Australia
  - Paincare Perth, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: No